CLINICAL TRIAL: NCT03834454
Title: How Low Can we go: A Double-blinded Randomized Controlled Trial to Compare Bupivacaine 5 mg and Bupivacaine 7.5 mg for Spinal Anesthesia in Cesarian Delivery in Indonesian Population
Brief Title: Bupivacaine 5 mg vs 7.5 mg for Spinal Anesthesia in Cesarean Delivery in Indonesian Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Susilo Chandra, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes027
Record Dates: First submitted 2019-02-01; First posted 2019-02-08 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Cesarean Section; Hypotension Drug-Induced; Spinal Anesthesia; Postoperative Complications
Keywords: pregnancy; caesarean section; spinal anesthesia; bupivacaine; opioid; hypotension; intraoperative; postoperative
MeSH Terms: conditions — Hypotension; Postoperative Complications | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Simple randomization will be conducted using a software by one of the researchers (HA) into two groups with equal size. To ensure the concealment, the randomization list will be kept in a sealed enveloped and opened by the physician who administered the spinal anesthesia just before the surgery. Data recording will be conducted by independent observers. This is a double-blinded study for the subjects and for the observers. The enrollment of the participants will be conducted by HA. Patients will not be notified about the dose scheme. Physician who performed the spinal anesthesia are different from the observers. Observers are junior residents trained to test the spinal adequacy and to perform monitoring in spinal anesthesia. It us not possible to blind the physicians who perform the spinal anesthesia because they will notice the volume difference.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine 5 mg (Active Comparator): 5 mg hyperbaric bupivacaine 0.5% and 25 mcg fentanyl for spinal anesthesia
  Interventions: Drug: Bupivacaine
- Bupivacaine 7.5 mg (Active Comparator): 7.5 mg hyperbaric bupivacaine 0.5% and 25 mcg fentanyl for spinal anesthesia
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — 5 mg hyperbaric bupivacaine 0.5% and 25 mcg fentanyl for spinal anesthesia
  Other Names: 5 mg hyperbaric bupivacaine 0.5%
  Arms: Bupivacaine 5 mg
Drug: Bupivacaine — 7.5 mg hyperbaric bupivacaine 0.5% and 25 mcg fentanyl for spinal anesthesia
  Other Names: 7.5 mg hyperbaric bupivacaine 0.5%
  Arms: Bupivacaine 7.5 mg

SUMMARY:
This study aims to evaluate the efficacy of hyperbaric 5 mg bupivacaine + fentanyl 25 mcg versus hyperbaric 7.5 mg bupivacaine + fentanyl 25 mcg to lower incidence of hypotension

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects will be recruited using consecutive sampling method. Sample size was determined using alpha 5%, power 80%, and the difference of the incidence of hypotension 20%. The sample of each group is 56 patients. The investigators will use ECG, blood pressure monitoring, and pulse oxymetry for the standard monitoring. Patients will be given oxygen 3 L/minute via nasal cannula. Before the spinal anesthesia, patients will be given co-loading 500 ml of Ringer Lactate. Patients will be in sitting position while the lumbal puncture is conducted using 27G Quincke in the level of L3-4 or L4-5 or Tuffier's line. After ensuring that the tip of the needle is in the subarachnoid space, the drug will be administered with the speed of 0.2 mL/s. All the procedure will be conducted in sterile condition. Patients will receive ketoprofen suppositoria as the postoperative analgesia and can be discharged to the ward when the Aldrete's score is more than 8.

The onset of sensoric blockade is assessed using pinprick test until the level of T6 or maximum until 20 minute. The peak value will be recorded. The motor blockade will be assessed using the Bromage scale. Incision will be done when the level of sensory block reached T6. If patients report pain after delivery of the baby, intravenous fentanyl 0,67-1 mcg/kg will be given twice with the interval of 10 minutes. If pain persists, conversion to general anesthesia will be conducted.

The measurement of blood pressure, heart rate, respiratory rate, temperature, and O2 saturation will be recorded during the minute of 3, 6, 9, 12, 15, 20, 30, 40, 50, and 60 after the spinal anesthesia is administered or until the baby is delivered. Patients will be recorded as hypotensive when she experienced reduction of blood pressure more than 30% from baseline or systolic pressure less than 100 mmHg from the moment the spinal anesthesia is administered until the baby is delivered. If the systolic pressure is less than 90 mmHg, patient will be given ephedrine 5 mg iv that is repeated every minute until the systolic pressure is over 90 mmHg.

The duration of the surgery is also recorded. Nausea, vomiting, syncope, dizziness, chest discomfort, and other intraoperative complaint will be recorded. Postoperative nausea and vomiting, itching, shivering, back pain, Post Dural Puncture Headache (PDPH), and Transient Neurologic Symptoms (TNS) will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with ASA PS 1-3
* age 18-40 years old
* in an elective or emergency cesarean delivery using spinal anesthesia

Exclusion Criteria:

* patients with contraindication of spinal anesthesia
* have history of allergy to bupivacaine or fentanyl
* with eclampsia
* valvular heart disease
* congenital heart disease
* coronary heart disease
* twin pregnancy
* morbid obesity (BMI >=40)
* pre-partum hemorrhage with hemodynamic instability

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 112 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension | 60 minutes
  recorded during the minute of 3, 6, 9, 12, 15, 20, 30, 40, 50, and 60 after the spinal anesthesia will be administered or until the baby is delivered

SECONDARY OUTCOMES:
Adequacy of Anesthesia | 120 minutes
  Requirement of additional local anesthetics
Quality of anesthesia: as reported by patients and surgeons | 120 minutes
  Quality of anesthesia as reported by patients and surgeons
Motor recovery | 10 hours
  Duration of motor recovery after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arzola C, Wieczorek PM. Efficacy of low-dose bupivacaine in spinal anaesthesia for Caesarean delivery: systematic review and meta-analysis. Br J Anaesth. 2011 Sep;107(3):308-18. doi: 10.1093/bja/aer200. Epub 2011 Jul 14. PMID 21764820
- [Background] Rollins M, Lucero J. Overview of anesthetic considerations for Cesarean delivery. Br Med Bull. 2012;101:105-25. doi: 10.1093/bmb/ldr050. Epub 2012 Jan 4. PMID 22219238
- [Background] Lee A, Ngan Kee WD, Gin T. Prophylactic ephedrine prevents hypotension during spinal anesthesia for Cesarean delivery but does not improve neonatal outcome: a quantitative systematic review. Can J Anaesth. 2002 Jun-Jul;49(6):588-99. doi: 10.1007/BF03017387. PMID 12067872
- [Background] Banerjee A, Stocche RM, Angle P, Halpern SH. Preload or coload for spinal anesthesia for elective Cesarean delivery: a meta-analysis. Can J Anaesth. 2010 Jan;57(1):24-31. doi: 10.1007/s12630-009-9206-7. Epub 2009 Oct 27. PMID 19859776
- [Background] Practice Guidelines for Obstetric Anesthesia: An Updated Report by the American Society of Anesthesiologists Task Force on Obstetric Anesthesia and the Society for Obstetric Anesthesia and Perinatology. Anesthesiology. 2016 Feb;124(2):270-300. doi: 10.1097/ALN.0000000000000935. No abstract available. PMID 26580836
- [Background] Qiu MT, Lin FQ, Fu SK, Zhang HB, Li HH, Zhang LM, Li Q. Combination of low-dose bupivacaine and opioids provides satisfactory analgesia with less intraoperative hypotension for spinal anesthesia in cesarean section. CNS Neurosci Ther. 2012 May;18(5):426-32. doi: 10.1111/j.1755-5949.2012.00306.x. PMID 22533726
- [Background] Ituk U, Habib AS. Enhanced recovery after cesarean delivery. F1000Res. 2018 Apr 27;7:F1000 Faculty Rev-513. doi: 10.12688/f1000research.13895.1. eCollection 2018. PMID 29770203
- [Background] Corso E, Hind D, Beever D, Fuller G, Wilson MJ, Wrench IJ, Chambers D. Enhanced recovery after elective caesarean: a rapid review of clinical protocols, and an umbrella review of systematic reviews. BMC Pregnancy Childbirth. 2017 Mar 20;17(1):91. doi: 10.1186/s12884-017-1265-0. PMID 28320342
- [Background] Leo S, Sng BL, Lim Y, Sia AT. A randomized comparison of low doses of hyperbaric bupivacaine in combined spinal-epidural anesthesia for cesarean delivery. Anesth Analg. 2009 Nov;109(5):1600-5. doi: 10.1213/ANE.0b013e3181b72d35. PMID 19843797
- [Background] Ben-David B, Miller G, Gavriel R, Gurevitch A. Low-dose bupivacaine-fentanyl spinal anesthesia for cesarean delivery. Reg Anesth Pain Med. 2000 May-Jun;25(3):235-9. PMID 10834776
- [Background] Ota E, Haruna M, Suzuki M, Anh DD, Tho le H, Tam NT, Thiem VD, Anh NT, Isozaki M, Shibuya K, Ariyoshi K, Murashima S, Moriuchi H, Yanai H. Maternal body mass index and gestational weight gain and their association with perinatal outcomes in Viet Nam. Bull World Health Organ. 2011 Feb 1;89(2):127-36. doi: 10.2471/BLT.10.077982. Epub 2010 Nov 10. PMID 21346924